CLINICAL TRIAL: NCT05907902
Title: Aspirin Treatment for Small Unruptured InTracranial Aneurysms With Ischemic cereBrovascuLar diseasE (AT-SUITABLE): a Phase 3, Multicenter, Prospective, Randomized, Open-label, Blinded-endpoint Controlled Trial
Brief Title: Aspirin Treatment for Small Unruptured InTracranial Aneurysms With Ischemic cereBrovascuLar diseasE
Acronym: AT-SUITABLE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Dr. Yong Cao, deputy director, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-I2M-C&T-B-114
Record Dates: First submitted 2023-05-22; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Intracranial Aneurysm; Cerebrovascular Disease
Keywords: Intracranial Aneurysm; Cerebrovascular Diseases; ischemic cerebrovascular disease; aspirin; Randomized Controlled Trial
MeSH Terms: conditions — Intracranial Aneurysm; Cerebrovascular Disorders

STUDY DESIGN:
Intervention Model Description: Participants are assigned to two groups in parallel for the duration of the study.
Who Masked: Outcomes Assessor
Masking Description: blinded-endpoint, PROBE design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin (Experimental): low-dose aspirin, 100 mg once daily, one 100mg tablet
  Interventions: Drug: Aspirin Enteric-coated Tablets
- standard protocol (No Intervention): standard of care, UIA management according to guidelines.

INTERVENTIONS:
Drug: Aspirin Enteric-coated Tablets — low-dose aspirin 100 mg once daily (one 100mg tablet).
  Other Names: Bayer
  Arms: Aspirin

SUMMARY:
The management of small unruptured intracranial aneurysms (UIA) with ischemic cerebrovascular disease (ICVD) has been a very controversial topic in neurosurgery. Thus, we initiated a multicenter, prospective, randomized controlled trial (PROBE) design to elucidate in UIA patients with ICVD who do not qualify for preventive endovascular or neurosurgical intervention whether aspirin treatment decreases the risk of aneurysm growth and rupture.

DETAILED DESCRIPTION:
Unruptured IAs are prevalent cerebrovascular disorders affecting approximately 3%-5% of the general population. The mortality rate associated with the rupture of UIAs stands at around 30%-40%, with over one-third of survivors experiencing significant neurological deficits. Currently, there are no established guidelines for the management of UIAs with ICVD. Our AIUIA trial is the inaugural randomized study investigating the potential of an anti-inflammatory strategy in mitigating aneurysm growth or rupture in patients with UIAs and ICVD who do not undergo preventive occlusion. It has the potential to provide level-A evidence that supports the aforementioned patient management approach.

ELIGIBILITY:
Inclusion Criteria:

* patients aged more than 18 and less than 80 years
* patients with UIAs < 5 and ≥2 mm in the greatest diameter confirmed by MR angiography (MRA), computed tomography angiography (CTA) , or digital subtraction angiography (DSA)
* patients with either symptomatic ICVD (ischemic stroke or transient ischemic attack) or asymptomatic ICVD (clinically silent lacunar infarction identified on brain CT/MR imaging)
* last aneurysm imaging with either CTA or MRA or DSA within the last 3 months
* ability of the subject to understand character and individual consequences of clinical trial
* patients who provided written informed consent
* patients who consented to follow-up imaging with the same MR angiography or CT angiography modality

Exclusion Criteria:

* multiple aneurysms
* a history of intracranial aneurysm rupture-related hemorrhage
* a family history of intracranial aneurysm
* a history of vascular malformation (brain arteriovenous malformation, moyamoya disease, arteriovenous fistula, etc.), brain tumor, hydrocephalus, or hypertensive cerebral hemorrhage etc.
* MR contraindications (metallic implant, contrast medium allergy, claustrophobia, etc).
* a precondition modified Rankin Scale (mRS) score > 2
* fusiform or daughter sac UIAs
* an allergy to aspirin
* other contraindications for aspirin not yet mentioned, in the dosage of 100 mg/day (e.g. bleeding disorders, gastric or intestinal ulcers, acute liver failure or kidney failure, severe heart failure, treatment with methotrexate in a dosage 15 mg/week or above)
* pregnancy and lactation
* participation in another clinical trial or observation period of competing trials
* residence in a rural area that prevented regular follow-up
* poor compliance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 824 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
number of participants with aneurysm rupture or growth | 24 months
  primary composite outcome involving aneurysm growth ((1) ≥1.0mm in at least 1 direction by identical imaging modalities, (2) ≥0.5 mm in 2 directions by identical imaging modalities, and (3) an indisputable change in aneurysm shape) or rupture on repeated magnetic resonance- or CT-angiography within 24 months after randomization.

SECONDARY OUTCOMES:
number of participants with aneurysm rupture | 24 months
  Individual components of the primary composite outcome, aneurysm rupture within 24 months after randomization.
number of participants with aneurysm growth on repeated angiography | 24 months
  Individual components of the primary composite outcome, aneurysm growth ((1) ≥1.0mm in at least 1 direction by identical imaging modalities, (2) ≥0.5 mm in 2 directions by identical imaging modalities, and (3) an indisputable change in aneurysm shape) on repeated magnetic resonance- or CT-angiography or DSA within 24 months after randomization.
degree of C-reaction protein level change | 24 months
  change of inflammatory biomarkers, serum C-reaction protein level
degree of cytokines level change | 24 months
  change of inflammatory biomarkers, cytokines including TNF-α, IL-6, IL-8, IL-10, IL-1β, IL-2R etc.
recurrent or new ischemic events | 24 months
  the incidence of recurrent or new ischemic events (symptoms suggestive of ischemic stroke or transient ischemic attack (TIA) and confirmed by neurologists in the town/village clinic of their choice)
any hemorrhagic stroke | 24 months
  the incidence of any hemorrhagic stroke, defined as the acute extravasation of blood into the brain parenchyma or subarachnoid space with associated neurological symptoms and a bleeding area far from the aneurysm location
any systematic bleeding | 24 months
  the incidence of systematic bleeding
all cause mortality | 24 months
  rate of overall mortality
number of participants with de novo aneurysm on repeated angiography | 24 months
  development of de novo aneurysm on serial imaging
adverse events (AEs)/serious adverse events (SAEs) | 24 months
  all adverse and serious adverse events pertaining to the aspirin

CONTACTS AND LOCATIONS:
Overall Officials: Yong Cao, MD, Principal Investigator — Department of Neurosurgery, Beijing Tiantan Hospital, Capital Medical University
Locations (2):
- China (2):
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Result] Weng JC, Wang J, Du X, Li H, Jiao YM, Fu WL, Huo R, Yan ZH, Xu HY, Wang S, Cao Y, Zhao JZ; Small Unruptured Aneurysms Study Group. Safety of Aspirin Use in Patients With Stroke and Small Unruptured Aneurysms. Neurology. 2021 Jan 5;96(1):e19-e29. doi: 10.1212/WNL.0000000000010997. Epub 2020 Oct 14. PMID 33055274
- [Result] Weng JC, Wang J, Li H, Jiao YM, Fu WL, Huo R, Yan ZH, Xu HY, Zhan J, Wang S, Du X, Cao Y, Zhao JZ; Small Unruptured Aneurysms Study Group. Aspirin and Growth of Small Unruptured Intracranial Aneurysm: Results of a Prospective Cohort Study. Stroke. 2020 Oct;51(10):3045-3054. doi: 10.1161/STROKEAHA.120.029967. Epub 2020 Sep 3. PMID 32878566